CLINICAL TRIAL: NCT03762057
Title: Prevalence, Risk Factors, and Prognostic Factors of Intraabdominal Hypertension and Abdominal Compartment Syndrome in Critically Ill Surgical Patients in Ramathibodi Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Cherdkiat karnjanarachata, MD, Ramathibodi Hospital
Other Study IDs: CK999
Record Dates: First submitted 2018-11-30; First posted 2018-12-03 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Intraabdominal Hypertension; Abdominal Compartment Syndrome
Keywords: Intraabdominal Hypertension; Abdominal Compartment Syndrome; Prevalence; Risk factors; ICU; Surgical
MeSH Terms: conditions — Intra-Abdominal Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical patients: All postoperative patients admitted to surgical ICU with foley catheter in place
  Interventions: Diagnostic Test: Intraabdominal pressure monitoring

INTERVENTIONS:
Diagnostic Test: Intraabdominal pressure monitoring — Classic manometry technique measurement once daily

SUMMARY:
To identified prevalence, risk factors, and prognostic factors of IAH and ACS in surgical critically ill patients in institutional hospital

DETAILED DESCRIPTION:
Every postoperative patients admitted to surgical ICU who meet inclusion criteria will be asked for informed consent. After obtained, intraabdominal pressure (IAP) will be measured through already placed Foley's catheter simultaneously with patients's data record. If patients don't have IAH or ICS, IAP will be measured daily until discharge from ICU or removal of Foley's catheter. If patients have IAH or ACS, IAP will be measured every 6-8 hours until IAP is less than 12 mmHg then it will be measures daily until discharge from ICU or removal of Foley's catheter. After completion of data collection, data will be analyzed accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Postoperative patient admitted to surgical ICU
* Age >/= 18
* Foley's catheter in place

Exclusion Criteria:

* Patient refusal
* Underwent neo-bladder procedure
* Need continuous bladder irrigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All postoperative adult patients admitted to institutional surgical ICUs.
Sampling Method: Non-Probability Sample
Enrollment: 303 (Estimated)
Dates: Start 2018-12-10 (Estimated); Primary Completion 2019-12-10 (Estimated); Study Completion 2020-06-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of intraabdominal hypertension and abdominal compartment syndrome | Within 30 days of ICU admission
  Prevalence of intraabdominal hypertension and abdominal compartment syndrome

SECONDARY OUTCOMES:
Risk factors of intraabdominal hypertension and abdominal compartment syndrome | Within 30 days of ICU admission
  Risk factors of intraabdominal hypertension and abdominal compartment syndrome
Prognostic factors of death after developing intraabdominal hypertension and abdominal compartment syndrome | Within 30 days of ICU admission
  Prognostic factors of death after developing intraabdominal hypertension and abdominal compartment syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Cherdkiat Karnjanarachata, MD, Principal Investigator — Faculty of medicine, Ramathibodi Hospital
Locations (1):
- Ramathibodi Hospital, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No